CLINICAL TRIAL: NCT01750437
Title: Randomized, Double-blind, Active-controlled, Multi-center Phase 2 Clinical Trial to Investigate the Safety, Tolerability and Efficacy of YH1885L in Patients With Non-erosive Reflux Disease(NERD)
Brief Title: Phase 2 Clinical Trial to Investigate the Safety, Tolerability and Efficacy of YH1885L in Patients With Non-erosive Reflux Disease(NERD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YH1885L-201
Record Dates: First submitted 2012-12-12; First posted 2012-12-17 (Estimated); Last update posted 2014-07-10 (Estimated); Status verified 2014-07

CONDITIONS: Non-erosive Reflux Disease
Keywords: NERD
MeSH Terms: conditions — Non-Erosive Reflux Disease | interventions — Esomeprazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- YH1885L 33.3 mg (Experimental): TID, Subject takes it for 4 week.
  Interventions: Drug: YH1885L(Revaprazan)
- YH1885L 50mg (Experimental): BID, Subject takes it for 4 week.
  Interventions: Drug: YH1885L(Revaprazan); Drug: placebo
- YH1885L 66.6 mg (Experimental): TID, Subject takes it for 4 week.
  Interventions: Drug: YH1885L(Revaprazan)
- YH1885L 100mg (Experimental): BID, Subject takes it for 4 week.
  Interventions: Drug: YH1885L(Revaprazan); Drug: placebo
- Esomeprazole 20mg (Active Comparator): QD, Subject takes it for 4 week.
  Interventions: Drug: Esomeprazole 20mg; Drug: placebo

INTERVENTIONS:
Drug: YH1885L(Revaprazan)
  Arms: YH1885L 100mg; YH1885L 33.3 mg; YH1885L 50mg; YH1885L 66.6 mg
Drug: Esomeprazole 20mg
  Other Names: Nexium
  Arms: Esomeprazole 20mg
Drug: placebo
  Arms: Esomeprazole 20mg; YH1885L 100mg; YH1885L 50mg

SUMMARY:
Randomized, double-blind, active-controlled, multi-center phase 2 clinical trial to investigate the safety, tolerability and efficacy of YH1885L in patients with non-erosive reflux disease(NERD)

ELIGIBILITY:
Inclusion Criteria:

* subjects who signed written informed consent form
* more than 20 yr subject
* subjects who agree the use of medically accepted birth control during trial
* grade N, M by EGD test
* subject who experience 2 day out of 1 week during recent 1 month
* subject who experience 2 day out of 1 week during run-in period

Exclusion Criteria:

* subjects who can write the diary by himself, herself
* pregnant woman, breastfeeding woman
* allgeric or intolerabiliy to revaprazan or esomeprazole
* feeling of heavy stomach, distention
* surgery history in stomach or esophagus
* active medical history of stomach, esophagus area
* other system disorder which can disturb this trial
* Hep B, C virus, HIV carrier or patients
* past history of malignant tumor
* any psychiatric past or current history
* abnormal lab test
* abnormal ecg test
* zollinger-ellison disease
* current or past history of substance, drug abuse
* subject who should regulary takes medication which can disturb this trial

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2013-01; Primary Completion 2013-10 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
the rate of subject who had 'complete recovery' of symptom after 4 week administration | 4 week
  'complete recovery' means subjects never experience heartburn or acid regurgitation during last 1 week.

SECONDARY OUTCOMES:
the rate of subject who had 'appropriate recovery' of symptom after 4 week administration | 4 week
  'Appropriate recovery' means subjects experience heartburn or acid regurgitation only 1 or less during last 1 week.
the rate of subject who had 'complete recovery' after 1 week, 2 week, 3 week IP administraion | 3 week
the rate of subject who had 'appropriate recovery' after 1 week, 2 week, 3 week IP administraion | 3 week
the number of night symptom-free day after IP administration | 1 week, 2 week, 3 week, 4 week
  Symptoms means "Heartburn or Acid regurgitation"
the rate of subjects who have reduced average symptom score(more than 1) comparing to baseline score | 1 week, 2 week, 3 week, 4 week
Evalution of Clinical Global Impression of Change | 4 week
Evaluation of Patient Global Impression of Change | 4 week
the change of SF-36 Survey score between baseline and completion visit | 4 week
the change of ESS survey score among baseline, 2 week and 4 week | 2, 4 week
  ESS stands for Epworth sleepiness scale.
Safety | 4 week
  AE, Physical exam, 12-lead ECG, Vital signs, laboratory test

OTHER OUTCOMES:
Comparison of H.pylori(+),(-) subjects about primay and seconday outcome | 4 week

CONTACTS AND LOCATIONS:
Locations (10):
- South Korea (10):
  - Catholic yeouido sungmo hospital, Seoul, Seoul
  - DongA university hospital, Busan
  - Kyungbook University hospital, Daegu
  - Chungnam university hospital, Daejeon
  - Catholic Incheon hospital, Incheon
  - Jeonbuk University hospital, Jeonju
  - Asan hospital, Seoul
  - Konkuk unversity hospital, Seoul
  - Kyunghee university hospital, Seoul
  - Seoul university hospital, Seoul